CLINICAL TRIAL: NCT05838339
Title: Are You Daydreaming? Co-creation to Promote Healthy Sleep in Adolescents in a School Context: a Health CASCADE Protocol
Brief Title: Are You Daydreaming?
Acronym: Health CASCADE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ONZ-2022-0174
Record Dates: First submitted 2022-11-07; First posted 2023-05-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-06

CONDITIONS: Sleep Hygiene; Sleep; Poor Quality Sleep
Keywords: Adolescence; Sleeping behavior; Co-creation; School-based intervention; School staff; Parents; Mental Health; Sleep; Motivation; Ownership; Health Promotion
MeSH Terms: conditions — Sleep Hygiene; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The investigators aim to conduct a pilot three-arm controlled trial with a mixed methods approach. Schools will be assigned to one of three groups: 1) co-creation intervention group (shortened co-creation process), 2) standard implementation group (no co-creation process), and 3) control group. After the implementation of the intervention, effect and process will be evaluated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Co-creation School (Experimental): An existing healthy sleep intervention will be scaled up using a shortened co-creation process. An effect- and process evaluation will be performed.
  Interventions: Behavioral: Healthy Sleep Intervention
- Standard Implementation School (Active Comparator): The existing healthy sleep intervention will be implemented without using a co-creation approach. An effect- and process evaluation will be performed.
  Interventions: Behavioral: Healthy Sleep Intervention
- Control School (No Intervention): No intervention will be implemented. An effect evaluation will be performed.

INTERVENTIONS:
Behavioral: Healthy Sleep Intervention — The existing intervention consists of the following components: Posters, Instagram, kick-off event, flyer for parents, parents-teacher conference, class discussions, app, classes on sleep (and relaxation), blue lights installations, alarm clocks and t-shirts, T-days without phone in the bedroom (Tuesdays and Thursdays), class competition.
  Arms: Co-creation School; Standard Implementation School

SUMMARY:
Health CASCADE (Marie Skłodowska-Curie grant agreement n° 956501) aims to address complex public health problems by making co-creation a scientifically sound methodology, aided by evidence-based methods, practices, and technologies. The current study, which focuses on co-creation in the school context is part of this overarching European project.

Healthy sleep is important for adolescents' mental and physical health and cognitive functioning. However, sleep difficulties are among the top three health complaints in European adolescents. This indicates a need for successful interventions.

Co-creation is a promising approach to design tailored interventions. By actively involving all relevant stakeholders, co-creation has been shown to increase self-efficacy, self-consciousness, empowerment, and feelings of ownership. However, co-created interventions are localized and therefore less generalizable to a broader population. Moreover, the process is very time- and cost- consuming. To make co-creation more feasible, research should focus on the upscaling of existing interventions. The investigators propose that the co-creation process is still absolutely vital for intervention success but that it can be shortened.

The investigators aim to scale up an existing intervention to promote healthy sleep. This existing intervention was developed using co-creation together with the target group (adolescents aged 13 to 15) and parents, and implemented with support of teachers and fellow students. To investigate whether the shorter co-creation process is needed in order to scale up the intervention to another setting and context, the investigators will use a three-arm cluster controlled trial. This will include one co-creation intervention school, one standard implementation school (this school receives the existing intervention without a shortened co-creation process), and one control school. The co-creation process will be structured by using the Intervention Mapping Protocol to ensure an evidence-based framework. The effect of the intervention will be evaluated using actigraphy and questionnaires, while the process will be evaluated using questionnaires, interviews, and focus groups.

DETAILED DESCRIPTION:
The aim of this study is to scale up an existing sleep intervention (co-created with adolescents and parents, and implemented with the support of teachers and fellow students) in Flanders to improve sleeping behavior. Scaling up an intervention is defined as transferring an intervention to another context, setting, and group. As co-created interventions are localized by nature, the researchers will investigate whether this existing intervention can be scaled up to a new context, setting, and group while the aim of the intervention remains the same, i.e., improving healthy sleeping behavior in adolescents. To test this, a co-creation school, standard implementation school, and control school will be recruited. Below, the investigators will describe what will be expected from each condition.

Co-creation school: Scaling up the existing sleep intervention to a new context, setting, and group will proceed in the co-creation school. The existing intervention will be adapted to the culture of this school, based on students', school staff's, and parents' perspective on the health problem (unhealthy sleeping behavior in adolescents) and thoughts on the components of the existing intervention. To adapt the existing sleep intervention, action groups will be composed. Every action group contains a maximum of 10 individuals.

* Action group adolescents: This action group consists of a maximum of 10 students from the 6th and 7th grade (1st grade secondary school, Belgian school system). The participants will be involved in the adaptation of existing intervention components. Furthermore, participants will implement the adapted intervention at school.
* Action group school staff: This action group consists of a maximum of 10 individuals working at the co-creation school. Participants will be involved in designing an implementation plan for the intervention. Moreover, participants will be asked to check the adapted components for feasibility.
* Action group parents: This action group consists of a maximum of 10 parents who have at least one child in the 6th or 7th grade of the co-creation school. Parents will be involved in the adaptation of the parental intervention components of the existing intervention.
* Co-facilitators: Students of the 12th grade (year 6 secondary school, Belgian school system) will be involved as co-facilitators. This means that the students of the 12th grade will facilitate the co-creation sessions designed for the students of the 6th and 7th grade together with the researchers.

Standard implementation school: To test the added value of the shortened co-creation process and to show that this process is needed to build ownership and empowerment, the existing sleep intervention will be implemented without the shortened co-creation process. The standard implementation school will be provided with a manual and a training about the implementation of the intervention.

Control school: To test the overall effect of the intervention a control group is needed. None of the interventions will be implemented at the control school and therefore the school staff do not have to take part in the measurements.

In total, the intervention in both the co-creation school and the standard implementation school will take 9 weeks.

Effect evaluation: To test the effect of the intervention, students (n = 378, based on a power analysis performed in R) will be invited to take part in three measurements (baseline, posttest (after the intervention), and follow-up (sixth months after the end of the intervention)) in all three arms. For members of the action group, a fourth measure will be administered (in-between baseline and posttest) to investigate whether the co-creation process itself can lead to changes in specific variables (see measures section). In order to compare the co-creation process to a standard implementation training, this fourth measurement will also be assessed among individuals involved in the implementation in the standard implementation school. To objectively measure sleep, participants will be asked to wear a GENEActiv device for 7 consecutive days at each of the three measurement points. Furthermore, participants will be invited to complete a questionnaire. This questionnaire will consist of questions about sleep duration, sleep quality, daytime sleepiness, sleep hygiene, determinants of sleeping behavior (knowledge, attitude, self-efficacy specifically related to sleeping behavior, social influence and social support, barriers), mental wellbeing, and feelings of empowerment and ownership. Furthermore, SES, puberty, and BMI will be assessed as important covariates. For students who are part of the action group (in the co-creation school) the questionnaire will also contain questions about general self-efficacy, and self-esteem. Moreover, students who are part of the action group will be invited to complete the whole questionnaire at one additional time point, namely after the shortened co-creation process. This measurement will enable us to investigate whether students in the action group experience more general self-efficacy and feelings of self-esteem as a result of participation in the co-creation process. Parents (ideally n = 378, one parent of each participating student) will be invited to complete questionnaires at the same measurement points as the students in all three arms. Parents' questionnaire will contain questions about knowledge and attitude about sleep, whether parents impose bedtime rules on children or have other supportive strategies, and questions regarding self-efficacy in engaging in these supportive strategies. Completion of questionnaires for students will take about one lesson (40-50 minutes). For parents, completion will take about 15 minutes.

Process evaluation: To evaluate the co-creation process as well as the implementation of the intervention, the investigators will use questionnaires, interviews, and focus groups. Students and parents from the action group will be asked to provide a short evaluation after every co-creation session. More extensive evaluations (focus group) will take place half-way during the development of the intervention, once the adaptation of the intervention is finished, and after the implementation of the intervention is done. Fellow students and parents, who are not part of the action group will be asked to evaluate the implementation of the intervention as well, using a short questionnaire. Students will also be invited to take part in focus groups. School staff (co-creation arm and standard implementation arm) will be invited to complete a questionnaire measuring motivation, empowerment, barriers for implementation, and general knowledge about sleep at three time points (baseline, pre-implementation, and after the intervention). Completion of questionnaires for school staff will take about 30 minutes. Moreover, school staff will be invited to take part in focus groups as well. These will take place at the same time points as for the students. Focus groups will take around 50 minutes (one lesson).

ELIGIBILITY:
Inclusion Criteria:

* Students must be aged between 11 and 13 years. Parents must have at least one child in the 6th or 7th Grade of the participating school.

Exclusion Criteria:

* None

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 382 (Actual)
Dates: Start 2022-10-04 (Actual); Primary Completion 2023-11-24 (Actual); Study Completion 2023-11-24 (Actual)

PRIMARY OUTCOMES:
Sleep quantity school days | Baseline
  Will be assessed using the Munich Chronotype Questionnaire for Children (MCTQ). Sleep onset will be calculated by adding the time of trying to go to sleep (item 2) and the time it really takes to fall asleep (item 3). Then, sleep quantity will be computed by calculating the difference between sleep onset and the time of waking up (item 4).
Sleep quantity free days | Baseline
  Will be assessed using the Munich Chronotype Questionnaire for Children (MCTQ). Sleep onset will be calculated by adding the time of trying to go to sleep (item 2) and the time it really takes to fall asleep (item 3). Then, sleep quantity will be computed by calculating the difference between sleep onset and the time of waking up (item 4).
Sleep quantity school days | Pre-intervention, after the co-creation process
  Will be assessed using the Munich Chronotype Questionnaire for Children (MCTQ). Sleep onset will be calculated by adding the time of trying to go to sleep (item 2) and the time it really takes to fall asleep (item 3). Then, sleep quantity will be computed by calculating the difference between sleep onset and the time of waking up (item 4). The pre-intervention assessment will only be done for members of the action group.
Sleep quantity free days | Pre-intervention, after the co-creation process
  Will be assessed using the Munich Chronotype Questionnaire for Children (MCTQ). Sleep onset will be calculated by adding the time of trying to go to sleep (item 2) and the time it really takes to fall asleep (item 3). Then, sleep quantity will be computed by calculating the difference between sleep onset and the time of waking up (item 4). The pre-intervention assessment will only be done for members of the action group.
Sleep quantity school days | Immediately after the intervention
  Will be assessed using the Munich Chronotype Questionnaire for Children (MCTQ). Sleep onset will be calculated by adding the time of trying to go to sleep (item 2) and the time it really takes to fall asleep (item 3). Then, sleep quantity will be computed by calculating the difference between sleep onset and the time of waking up (item 4).
Sleep quantity free days | Immediately after the intervention
  Will be assessed using the Munich Chronotype Questionnaire for Children (MCTQ). Sleep onset will be calculated by adding the time of trying to go to sleep (item 2) and the time it really takes to fall asleep (item 3). Then, sleep quantity will be computed by calculating the difference between sleep onset and the time of waking up (item 4).
Sleep quantity school days | 6 months after the intervention
  Will be assessed using the Munich Chronotype Questionnaire for Children (MCTQ). Sleep onset will be calculated by adding the time of trying to go to sleep (item 2) and the time it really takes to fall asleep (item 3). Then, sleep quantity will be computed by calculating the difference between sleep onset and the time of waking up (item 4).
Sleep quantity free days | 6 months after the intervention
  Will be assessed using the Munich Chronotype Questionnaire for Children (MCTQ). Sleep onset will be calculated by adding the time of trying to go to sleep (item 2) and the time it really takes to fall asleep (item 3). Then, sleep quantity will be computed by calculating the difference between sleep onset and the time of waking up (item 4).
Objective sleep quantity school days | Baseline
  Will be assessed objectively using actigraphy (GENEActivs)
Objective sleep quantity free days | Baseline
  Will be assessed objectively using actigraphy (GENEActivs)
Objective sleep quantity school days | Pre-intervention, after the co-creation process
  Will be assessed objectively using actigraphy (GENEActivs). The pre-intervention assessment will only be done for members of the action group.
Objective sleep quantity free days | Pre-intervention, after the co-creation process
  Will be assessed objectively using actigraphy (GENEActivs). The pre-intervention assessment will only be done for members of the action group.
Objective sleep quantity school days | Immediately after the intervention
  Will be assessed objectively using actigraphy (GENEActivs)
Objective sleep quantity free days | Immediately after the intervention
  Will be assessed objectively using actigraphy (GENEActivs)
Objective sleep quantity school days | 6 months after the intervention
  Will be assessed objectively using actigraphy (GENEActivs)
Objective sleep quantity free days | 6 months after the intervention
  Will be assessed objectively using actigraphy (GENEActivs)
Sleep quality - general | Baseline
  Will be assessed using the short form of the Adolescent Sleep Wake Scale (s-ASWS)
Sleep quality - daytime sleepiness | Baseline
  Will be assessed using the Pediatric Daytime Sleepiness Scale (PDSS)
Sleep quality school days - SOL | Baseline
  Will be assessed with Sleep Onset Latency (SOL), item 3 of the MCTQ
Sleep quality free days - SOL | Baseline
  Will be assessed with Sleep Onset Latency (SOL), item 3 of the MCTQ
Objective sleep quality | Baseline
  Will be assessed objectively using actigraphy (GENEActivs)
Sleep quality - general | Pre-intervention, after the co-creation process
  Will be assessed using the short form of the Adolescent Sleep Wake Scale (s-ASWS). The pre-intervention assessment will only be done for members of the action group.
Sleep quality - daytime sleepiness | Pre-intervention, after the co-creation process
  Will be assessed using the Pediatric Daytime Sleepiness Scale (PDSS). The pre-intervention assessment will only be done for members of the action group.
Sleep quality school days - SOL | Pre-intervention, after the co-creation process
  Will be assessed with Sleep Onset Latency (SOL), item 3 of the MCTQ. The pre-intervention assessment will only be done for members of the action group.
Sleep quality free days - SOL | Pre-intervention, after the co-creation process
  Will be assessed with Sleep Onset Latency (SOL), item 3 of the MCTQ. The pre-intervention assessment will only be done for members of the action group.
Objective sleep quality | Pre-intervention, after the co-creation process
  Will be assessed objectively using actigraphy (GENEActivs). The pre-intervention assessment will only be done for members of the action group.
Sleep quality - general | Immediately after the intervention
  Will be assessed using the short form of the Adolescent Sleep Wake Scale (s-ASWS).
Sleep quality - daytime sleepiness | Immediately after the intervention
  Will be assessed using the Pediatric Daytime Sleepiness Scale (PDSS)
Sleep quality school days - SOL | Immediately after the intervention
  Will be assessed with Sleep Onset Latency (SOL), item 3 of the MCTQ
Sleep quality free days - SOL | Immediately after the intervention
  Will be assessed with Sleep Onset Latency (SOL), item 3 of the MCTQ
Objective sleep quality | Immediately after the intervention
  Will be assessed objectively using actigraphy (GENEActivs)
Sleep quality - general | 6 months after the intervention
  Will be assessed using the short form of the Adolescent Sleep Wake Scale (s-ASWS)
Sleep quality - daytime sleepiness | 6 months after the intervention
  Will be assessed using the Pediatric Daytime Sleepiness Scale
Sleep quality school days - SOL | 6 months after the intervention
  Will be assessed with Sleep Onset Latency (SOL), item 3 of the MCTQ
Sleep quality free days - SOL | 6 months after the intervention
  Will be assessed with Sleep Onset Latency (SOL), item 3 of the MCTQ
Objective sleep quality | 6 months after the intervention
  Will be assessed objectively using actigraphy (GENEActivs)

SECONDARY OUTCOMES:
Determinants of sleeping behavior | Baseline
  A questionnaire to assess psychosocial determinants of adolescents' sleeping behavior was developed. This questionnaire assesses knowledge, attitude, self-efficacy, social influence, barriers, and facilitators for healthy sleeping behavior, as well as sleep hygiene (nutrition, physical activity).
Determinants of sleeping behavior | Pre-intervention, after the co-creation process
  A questionnaire to assess psychosocial determinants of adolescents' sleeping behavior was developed. This questionnaire assesses knowledge, attitude, self-efficacy, social influence, barriers, and facilitators for healthy sleeping behavior, as well as sleep hygiene (nutrition, physical activity). The pre-intervention assessment will only be done for members of the action group.
Determinants of sleeping behavior | Immediately after the intervention
  A questionnaire to assess psychosocial determinants of adolescents' sleeping behavior was developed. This questionnaire assesses knowledge, attitude, self-efficacy, social influence, barriers, and facilitators for healthy sleeping behavior, as well as sleep hygiene (nutrition, physical activity).
Determinants of sleeping behavior | 6 months after the intervention
  A questionnaire to assess psychosocial determinants of adolescents' sleeping behavior was developed. This questionnaire assesses knowledge, attitude, self-efficacy, social influence, barriers, and facilitators for healthy sleeping behavior, as well as sleep hygiene (nutrition, physical activity).
Mental wellbeing | Baseline
  Mental wellbeing will be assessed with the Warwick Edinburgh Mental Wellbeing Scale (WEMWBS).
Mental wellbeing | Pre-intervention, after the co-creation process
  Mental wellbeing will be assessed with the Warwick Edinburgh Mental Wellbeing Scale (WEMWBS). The pre-intervention assessment will only be done for members of the action group.
Mental wellbeing | Immediately after the intervention
  Mental wellbeing will be assessed with the Warwick Edinburgh Mental Wellbeing Scale (WEMWBS).
Mental wellbeing | 6 months after the intervention
  Mental wellbeing will be assessed with the Warwick Edinburgh Mental Wellbeing Scale (WEMWBS).
Self-efficacy | Baseline
  General Self-efficacy Scale (GSE) will be used to assess self-efficacy in children who are part of the action group.
Self-efficacy | Pre-intervention, after the co-creation process
  General Self-efficacy Scale (GSE) will be used to assess self-efficacy in children who are part of the action group.
Self-efficacy | Immediately after the intervention
  General Self-efficacy Scale (GSE) will be used to assess self-efficacy in children who are part of the action group.
Self-efficacy | 6 months after the intervention
  General Self-efficacy Scale (GSE) will be used to assess self-efficacy in children who are part of the action group.
Empowerment | Baseline
  Empowerment will be measured with the policy control dimension of the Social Political Control Scale for Youth (SPCS-Y) in both students and school staff as this scale focuses specifically on the school context.
Empowerment | Pre-intervention, after the co-creation process
  Empowerment will be measured with the policy control dimension of the Social Political Control Scale for Youth (SPCS-Y) in both students and school staff as this scale focuses specifically on the school context. The pre-intervention assessment will only be done for members of the action group.
Empowerment | Immediately after the intervention
  Empowerment will be measured with the policy control dimension of the Social Political Control Scale for Youth (SPCS-Y) in both students and school staff as this scale focuses specifically on the school context.
Empowerment | 6 months after the intervention
  Empowerment will be measured with the policy control dimension of the Social Political Control Scale for Youth (SPCS-Y) in both students and school staff as this scale focuses specifically on the school context.
General motivation | Baseline
  The Dutch Basic Psychological Needs Satisfaction Needs Frustration Scale (BPNSFS) will be used to measure school staff's motivation.
General motivation | Pre-intervention, after the co-creation process
  The Dutch Basic Psychological Needs Satisfaction Needs Frustration Scale (BPNSFS) will be used to measure school staff's motivation.
General motivation | Immediately after the intervention
  The Dutch Basic Psychological Needs Satisfaction Needs Frustration Scale (BPNSFS) will be used to measure school staff's motivation.
Self-esteem | Baseline
  The Rosenberg Self-esteem Scale will be used to measure self-esteem in children who are part of the action group.
Self-esteem | Pre-intervention, after the co-creation process
  The Rosenberg Self-esteem Scale will be used to measure self-esteem in children who are part of the action group.
Self-esteem | Immediately after the intervention
  The Rosenberg Self-esteem Scale will be used to measure self-esteem in children who are part of the action group.
Self-esteem | 6 months after the intervention
  The Rosenberg Self-esteem Scale will be used to measure self-esteem in children who are part of the action group.
Motivation for implementation | Baseline
  The Motivation At Work Scale (MAWS) will be used to measure school staff's motivation for the implementation of the sleep intervention at school.
Motivation for implementation | Pre-intervention, after the co-creation process
  The Motivation At Work Scale (MAWS) will be used to measure school staff's motivation for the implementation of the sleep intervention at school.
Motivation for implementation | Immediately after the intervention
  The Motivation At Work Scale (MAWS) will be used to measure school staff's motivation for the implementation of the sleep intervention at school.
Barriers for implementation | Baseline
  Based on findings of previous research questions were formulated regarding certain barriers that can appear during the implemtation of a school-based intervention.
Barriers for implementation | Pre-intervention, after the co-creation process
  Based on findings of previous research questions were formulated regarding certain barriers that can appear during the implemtation of a school-based intervention.
Barriers for implementation | Immediately after the intervention
  Based on findings of previous research questions were formulated regarding certain barriers that can appear during the implemtation of a school-based intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Maïté Verloigne, Prof. dr., Principal Investigator — University Ghent
Locations (1):
- Ghent University, Ghent, East Flanders, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to share pseudonymized data within the Health CASCADE consortium and with fellow colleagues within the research group for secondary data analyses and teaching purposes. However, participants must re-consent for the use of their data in a new research project and domain.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data collection will take place from October 2022 until November 2023, afterwards data will be pseudonymised and shared. As Health CASCADE is a project that supports open science pseudonymised data will be available for the persons specified above forever.
Access Criteria: Everyone that possess the URL to the Zenodo Health CASCADE page can access the pseudonymized data files.
URL: https://zenodo.org/communities/health_cascade/

REFERENCES:
- [Background] Drake C, Nickel C, Burduvali E, Roth T, Jefferson C, Pietro B. The pediatric daytime sleepiness scale (PDSS): sleep habits and school outcomes in middle-school children. Sleep. 2003 Jun 15;26(4):455-8. PMID 12841372
- [Background] Leask CF, Sandlund M, Skelton DA, Altenburg TM, Cardon G, Chinapaw MJM, De Bourdeaudhuij I, Verloigne M, Chastin SFM; GrandStand, Safe Step and Teenage Girls on the Move Research Groups. Framework, principles and recommendations for utilising participatory methodologies in the co-creation and evaluation of public health interventions. Res Involv Engagem. 2019 Jan 9;5:2. doi: 10.1186/s40900-018-0136-9. eCollection 2019. PMID 30652027
- [Background] Roenneberg T, Keller LK, Fischer D, Matera JL, Vetter C, Winnebeck EC. Human activity and rest in situ. Methods Enzymol. 2015;552:257-83. doi: 10.1016/bs.mie.2014.11.028. Epub 2015 Jan 5. PMID 25707281
- [Background] Sufrinko AM, Valrie CR, Lanzo L, Bond KE, Trout KL, Ladd RE, Everhart DE. Empirical validation of a short version of the Adolescent Sleep-Wake Scale using a sample of ethnically diverse adolescents from an economically disadvantage community. Sleep Med. 2015 Oct;16(10):1204-6. doi: 10.1016/j.sleep.2015.07.002. Epub 2015 Jul 15. PMID 26429746
- [Background] Tennant R, Hiller L, Fishwick R, Platt S, Joseph S, Weich S, Parkinson J, Secker J, Stewart-Brown S. The Warwick-Edinburgh Mental Well-being Scale (WEMWBS): development and UK validation. Health Qual Life Outcomes. 2007 Nov 27;5:63. doi: 10.1186/1477-7525-5-63. PMID 18042300
- [Background] Vandendriessche A, Dierckens M, Delaruelle K, Deforche B. How Are Adolescents Sleeping? Conservative Estimates of Sleep Duration Underestimate the Problem. J Adolesc Health. 2021 Apr;68(4):830. doi: 10.1016/j.jadohealth.2020.12.137. No abstract available. PMID 33781473
- [Background] Wood C, Griffin M, Barton J, Sandercock G. Modification of the Rosenberg Scale to Assess Self-Esteem in Children. Front Public Health. 2021 Jun 17;9:655892. doi: 10.3389/fpubh.2021.655892. eCollection 2021. PMID 34222169
- [Background] Soenens, B., Sierens, E., Vansteenkiste, M., Dochy, F., & Goossens, L. (2012). Psychologically controlling teaching: Examining outcomes, antecedents, and mediators. Journal of Educational Psychology, 104(1), 108-120. https://doi.org/10.1037/a0025742
- [Background] Blais, M. R., Brière, N. M., Lachance, L., & Riddle, A. S. (1993). L'inventaire des motivations au travail de Blais. Revue québécoise de psychologie.
- [Derived] Delfmann LR, Vandendriessche A, de Boer J, Cardon G, Hunter SC, Dhondt K, Verloigne M, Deforche B. Co-adapting a healthy sleep intervention with adolescents: impact and process evaluation of a Health CASCADE pilot study. BMC Public Health. 2025 Nov 22;25(1):4411. doi: 10.1186/s12889-025-25412-2. PMID 41275198
- See also: Basic psychological need satisfaction need frustration scale — https://link.springer.com/article/10.1007/s11031-014-9450-1
- See also: General Self-efficacy Scale — http://userpage.fu-berlin.de/~health/selfscal.htm
- See also: Adolescent health and wellbeing — https://apps.who.int/iris/bitstream/handle/10665/332091/9789289055000-eng.pdf